CLINICAL TRIAL: NCT06071676
Title: Digital Versus Conventional Impression Used in The CAD / CAM Constructed 4- Implant Supported Mandibular Overdenture Base: Bone Height Changes
Brief Title: Digital Versus Conventional Impression CAD\CAM Constructed 4- Implant Supported Mandibular Overdenture Base
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M01010322
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2022-02

CONDITIONS: Implant Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional impression procedures (Other): Implant analogues were screwed to the transfer copings inside the impression and the master cast were obtained. Attachments were screwed to the analogues and metal housing wasplaced on their position on master cast. Master cast will be scanned extra orally to obtain STL file of the master cast.
  Interventions: Other: conventional impression group
- digital impression procedures (Other): A digital scanner (shining 3D scanner, Germany) was utilized to fabricate the definitive prostheses. The attachments were screwed to the implants intra orally and metal housing on their position which scanned by using intra oral scanner.
  * Intra oral scanner transformed into a virtual volume the three-dimensional geometry of dental arches using the principle of structured light. A scanning stitching strategy carried out by the same experienced investigator and applied to DIG group for the attachments on their position on implants.
  * The software automatically was applied a stitching algorithm in order to merge the two halves, based on the area between the two anterior implants, shared by both the separate scans.
  * The virtual model was created of the dental implant and attachments in position which used to obtain 3d printed master cast by using 3D printer (WANHAO desktop 3D printer, Zhejiang, China).
  Interventions: Other: digital impression group

INTERVENTIONS:
Other: conventional impression group — Silicon impression material loaded on plastic tray and inserted inside the patient mouth
  Arms: conventional impression procedures
Other: digital impression group — direct scanning was done using intraoral scanner to the female housing of the attachments on position
  Arms: digital impression procedures

SUMMARY:
This clinical study was done to compare between digital with conventional impression used in the CAD/CAM constructed 4- implant supported mandibular overdenture base regarding their effect on the bone height changes

DETAILED DESCRIPTION:
The patients were classified randomly into two equal groups according to impression techniques of mandibular implants and residual ridge:

Group 1: conventional impression group (CIG). Group 2: digital impression group (DIG).

For group 1 :

* Unscrew the provisional acrylic denture from the implants

  . - The long transfer copings (implant level) were screwed to the implants.
* The transfer copings were splinted with orthodontic ligature wire and light cure composite resin before impression making to prevent movement of the transfer coping during impression procedure.
* A stock/special tray was perforated to allow passing of the transfer copings through it without interference and permit unscrewing of the transfer after setting of the impression

  * - If there is large opening occurred, the opening was closed off using base plate wax to support the impression material, with the guide pins perforating the wax
  * - Inject the light body rubber base impression around the transfer coping. Fill the tray with a heavy body impression material and insert it intraorally till the tips of all the guide pins are appeared, clean the guide pin access holes from excess impression material.
* Unscrew the long transfer coping from the opining of the tray to allow it to be removed with the impression material.
* Implant analogues was screwed into the transfer coping.
* The impression was poured to obtain master cast then attachments(ball and socket attachments) were screwed to the implant analogues and metal housings placed on their position on master cast.
* The lower master cast was scanned using extra oral 3D scanner (DOF Swing dental scanner, Correa) to obtain the standard tessellation language (STL) file format.

For group 2 :

* A digital scanner (shining 3D scanner, Germany) was utilized to fabricate the definitive prostheses. The attachments were screwed to the implants intra orally and metal housing on their position which scanned by using intra oral scanner.
* Intra oral scanner transformed into a virtual volume the three-dimensional geometry of dental arches using the principle of structured light. A scanning stitching strategy carried out by the same experienced investigator and applied to DIG group for the attachments on their position on implants.
* IOS light source formerly kept parallel to the occlusal plane and started from the distal implant of the left quadrant and moved toward the anterior implant of the contralateral quadrant (right side); it was then moved back to the distal implant of the left side, tilting it toward the palatal side; the occlusal plane was crossed toward the buccal side and the camera moved again from the starting scanning point of the left side to the anterior implant of the right side trying to keep it perpendicular to the occlusal plane.
* The image was then inspected and missing regions were filled by fast passages of the camera over the related areas.
* The same scanning procedure was performed with the other half, from the anterior implant of the left quadrant to the distal implant of the contralateral quadrant (right side).
* The software automatically was applied a stitching algorithm in order to merge the two halves, based on the area between the two anterior implants, shared by both the separate scans.
* The virtual model was created of the dental implant and attachments in position which used to obtain 3d printed master cast by using 3D printer (WANHAO desktop 3D printer, Zhejiang, China).

Then for both groups

1. After approval of the virtual design preview of the permanent denture base by the investigator and technician, a pre polymerized denture base material (Ava Dent Digital Dental solutions HQ, Scottsdale, USA) were fabricated by CAD-CAM milling machine (DENTSPLY Sirona In Lab MC X5 laboratory milling machine, Germany) according to manufacturer' instructions.
2. The denture base was milled from Pre-polymerized CAD-CAM PMMA acrylic plates (98-mm diameter×25-mm thick) by using milling machine.
3. After the CAD-CAM permanent denture base milled, female parts (metal housing) of the attachments cemented on the prepared positions on the fitting surface of the denture base by using dual cure glass ionomer resin cement extra orally and cement excess removed from the lingual vents on the prepared positions of metal housing .
4. Record blocks were constructed on the master casts and used to record Maxillo-mandibular jaw relation by using milled permanent denture base.
5. Mounting of the maxillary cast was done on a semi-adjustable articulator† by the aid of maxillary face bow and the mandibular cast mounting was done in relation to the maxillary cast by centric inter occlusal wax wafer record.
6. Protrusive wax record was used for adjusting the horizontal condylar angle of the semi adjustable articulator, while the lateral condylar angle was adjusted according to Hanau equation: L = H / 8 + 12. Where H represents the horizontal condylar path inclination in degrees as established by a protrusive record and L represents the lateral condylar path inclination in degrees.
7. Maxillary anatomical and mandibular flat acrylic teeth‡ were arranged for lingualized balanced occlusion and try in was done in the patient's mouth.
8. For the lower permanent denture base teeth cemented on their positions by using self cure acrylic resin .
9. For the upper denture , flasking and processing was done into heat cured acrylic resin by the long curing cycle.
10. After finishing and polishing, the dentures were remounted to adjust any occlusal discrepancies and to ensure proper contact in centric and eccentric positions. Final adjustment of the occlusion was done intraorally.
11. The patient was instructed for proper insertion, removal, home care and hygiene and to use the denture until the evaluation session.

ELIGIBILITY:
Inclusion Criteria:

* All patient wearing maxillary conventional denture.
* All patients had temporary mandibular overdenture supported by vertically inserted 4-implant at least six months ago.
* A Cone Beam Computed Tomography (CBCT) done to verify the accurate position and success of the inserted implant.
* They were healthy, free from any systemic diseases relating to bone resorption such as uncontrolled diabetics or osteoporosis. This was achieved through medical history and clinical examination by physician.
* At least 15 mm restorative space must be available (from the mucosa covering the crest of the residual ridge to proposed occlusal plane) to permit construction of all types of tested prosthesis (class I according to Ahuja and Cagna). This was detected by a tentative jaw relation.
* All patients are of angel's class I maxillo-mandibular relationships.

Exclusion Criteria:

* Patients had head and neck radiotherapy, patients with bleeding disorders or hepatic patients.
* Patients with metabolic disorders as diabetes mellitus, osteoporosis and hepatic disorders that might affect osseointegration.
* Long term immunosuppress and corticosteroid drug therapy.
* Patient with abnormal habits as clenching and bruxism.
* Smoking patient.
* Uncooperative patients.
* Neuromuscular diseases.
* Patient with problems in TMJ.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Bone height changes | one year
  Long cone paralleling technique and a film holder designed specifically for implant imaging were used for intraoral radiograph. To maintain the same film- implant distance and cone implant distance, a modification was carried out for the film holder. This modification is a hole drilled exactly above the implant fixture so the distance was maintained during subsequent film exposures. A long screw of the impression coping was used to secure the holder to the implant. Through this modification, standardized radiographs were achieved.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed fouad, professor, Principal Investigator — specify Unaffiliated
Locations (1):
- Faculty of Dentistry, Al Mansurah, Egypt

REFERENCES:
- [Result] Goracci C, Franchi L, Vichi A, Ferrari M. Accuracy, reliability, and efficiency of intraoral scanners for full-arch impressions: a systematic review of the clinical evidence. Eur J Orthod. 2016 Aug;38(4):422-8. doi: 10.1093/ejo/cjv077. Epub 2015 Oct 20. PMID 26487391
- See also: Accuracy, reliability, and efficiency of intraoral scanners for full-arch impressions — https://pubmed.ncbi.nlm.nih.gov/26487391/